CLINICAL TRIAL: NCT02655471
Title: Effect of Raltegravir in Patients With Myelopathy/Tropical Spastic Paraparesis Associated With Infection by Human T-Lymphotropic Virus 1 (HTLV-1). Pilot Study
Brief Title: Effect of Raltegravir in Patients With Acute Tropical Spastic Paraparesis - Human T-Lymphotropic Virus 1 Infection
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 65384
Record Dates: First submitted 2015-11-16; First posted 2016-01-14 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: HTLV-I Infections; Tropical Spastic Paraparesis
MeSH Terms: conditions — HTLV-I Infections; Paraparesis, Tropical Spastic | interventions — Raltegravir Potassium; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HTLV-1 plus Tropical Spastic paraparesis (Experimental): Patients with recent onset of Tropical Spastic paraparesis due HTLV-1 will receive combination of "Raltegravir" and "Zidovudine" during 48 weeks
  Interventions: Drug: "Raltegravir" and "Zidovudine"

INTERVENTIONS:
Drug: "Raltegravir" and "Zidovudine" — Through measure of pro-viral load and clinical score, we evaluate about safety and efficacy of combination of Raltegravir 400 mg BID and zidovudine 300 mg BID in patients with recent onset of Tropical Spastic paraparesis due HTLV-1 during 48 weeks
  Other Names: "Raltegravir"; "Zidovudine"

SUMMARY:
This is a pilot study of intervention in a group of patients with tropical spastic paraparesis/ myelopathy to evaluate virologic and clinical response of raltegravir plus zidovudine in this group of patients.

DETAILED DESCRIPTION:
The study will the investigators develop in The Tropical Medicine Institute Alexander von Humboldt that is a referral center in Peru for diseases associated to Human T-Lymphotropic Virus 1 Infection (HTLV-1). The Institute has a cohort of around 600 patients currently being followed up and around 20 to 25 new patients are admitted every year with this disease.

This is a pilot study of intervention in a group of patients with tropical spastic paraparesis/ myelopathy to evaluate virologic and clinical response of raltegravir plus zidovudine in this group of patients on the follow-up of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* human t lymphotrophic virus 1 confirmed
* Tropical Spastic Paraparesis of recent onset (less than 4 years)

Exclusion Criteria:

* Pregnant or breastfeeding or unwilling to use contraception.
* Treatment with immunosuppressive, immunomodulatory or experimental treatments within the last 6 months of enrolment in the study.
* Patients presenting with medical disorder such as poorly controlled diabetes or arterial hypertension, severe cardiac insufficiency, unstable ischemic heart disease, abnormal liver function tests (>2.5 times upper limit normal (ULN)) and abnormal complete blood count (in particular leukopenia, as defined by a lymphocyte count <500, neutrophil <1.5 or platelet count < 100, or thrombocytopenia < 1.5 low limit normal (LLN), or any medical condition which, in the opinion of the chief investigator, would pose additional risk to the patient.
* Presence of human immunodeficiency virus antibodies.
* Patients with active hepatitis B or/and C with liver function tests >2.5 times ULN
* Exposure to any other investigational drug within 30 days of enrolment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Measure of proviral load | 48 weeks
  Evaluate the effect of raltegravir on proviral load , measured as copies/1000 PBMC, in patients with myelopathy of recent onset associated to HTLV-1 at 48 weeks.

SECONDARY OUTCOMES:
Measure of Disability Scale | 48 weeks
  Evaluate the effect of raltegravir on Kurtzke Expanded Disability Status Scale in patients with myelopathy of recent onset associated to HTLV-1 at 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Gotuzzo, MD, Principal Investigator — Instituto de Medicina Tropical Alexander von Humboldt; Fernando Mejía, MD, Principal Investigator — Instituto de Medicina Tropical Alexander von Humboldt
Locations (1):
- Instituto de Medicina Tropical Alexander von Humboldt, Lima, Peru

REFERENCES:
- [Result] Verdonck K, Gonzalez E, Van Dooren S, Vandamme AM, Vanham G, Gotuzzo E. Human T-lymphotropic virus 1: recent knowledge about an ancient infection. Lancet Infect Dis. 2007 Apr;7(4):266-81. doi: 10.1016/S1473-3099(07)70081-6. PMID 17376384
- [Result] Zurita S, Costa C, Watts D, Indacochea S, Campos P, Sanchez J, Gotuzzo E. Prevalence of human retroviral infection in Quillabamba and Cuzco, Peru: a new endemic area for human T cell lymphotropic virus type 1. Am J Trop Med Hyg. 1997 May;56(5):561-5. doi: 10.4269/ajtmh.1997.56.561. PMID 9180608
- [Result] Primo J, Siqueira I, Nascimento MC, Oliveira MF, Farre L, Carvalho EM, Bittencourt AL. High HTLV-1 proviral load, a marker for HTLV-1 associated myelopathy/tropical spastic paraparesis, is also detected in patients with infective dermatitis associated with HTLV-1. Braz J Med Biol Res. 2009 Aug;42(8):761-4. doi: 10.1590/s0100-879x2009005000008. Epub 2009 Jul 3. PMID 19578703
- [Result] Izumo S. Neuropathology of HTLV-1-associated myelopathy (HAM/TSP): The 50th Anniversary of Japanese Society of Neuropathology. Neuropathology. 2010 Oct;30(5):480-5. doi: 10.1111/j.1440-1789.2010.01135.x. PMID 20573027
- [Result] Varrin-Doyer M, Nicolle A, Marignier R, Cavagna S, Benetollo C, Wattel E, Giraudon P. Human T lymphotropic virus type 1 increases T lymphocyte migration by recruiting the cytoskeleton organizer CRMP2. J Immunol. 2012 Feb 1;188(3):1222-33. doi: 10.4049/jimmunol.1101562. Epub 2012 Jan 6. PMID 22227566
- [Result] Gill PS, Harrington W Jr, Kaplan MH, Ribeiro RC, Bennett JM, Liebman HA, Bernstein-Singer M, Espina BM, Cabral L, Allen S, et al. Treatment of adult T-cell leukemia-lymphoma with a combination of interferon alfa and zidovudine. N Engl J Med. 1995 Jun 29;332(26):1744-8. doi: 10.1056/NEJM199506293322603. PMID 7760890
- [Result] Hermine O, Allard I, Levy V, Arnulf B, Gessain A, Bazarbachi A; French ATL therapy group. A prospective phase II clinical trial with the use of zidovudine and interferon-alpha in the acute and lymphoma forms of adult T-cell leukemia/lymphoma. Hematol J. 2002;3(6):276-82. doi: 10.1038/sj.thj.6200195. PMID 12522449
- [Result] Seegulam ME, Ratner L. Integrase inhibitors effective against human T-cell leukemia virus type 1. Antimicrob Agents Chemother. 2011 May;55(5):2011-7. doi: 10.1128/AAC.01413-10. Epub 2011 Feb 22. PMID 21343468
- [Result] Trevino A, Parra P, Bar-Magen T, Garrido C, de Mendoza C, Soriano V. Antiviral effect of raltegravir on HTLV-1 carriers. J Antimicrob Chemother. 2012 Jan;67(1):218-21. doi: 10.1093/jac/dkr404. Epub 2011 Sep 29. PMID 21965433
- [Result] Gotuzzo E, Cabrera J, Deza L, Verdonck K, Vandamme AM, Cairampoma R, Vizcarra D, Cabada M, Narvarte G, De las Casas C. Clinical characteristics of patients in Peru with human T cell lymphotropic virus type 1-associated tropical spastic paraparesis. Clin Infect Dis. 2004 Oct 1;39(7):939-44. doi: 10.1086/423957. Epub 2004 Sep 1. PMID 15472843